CLINICAL TRIAL: NCT06709443
Title: Impact of Parental Presence on the Mean Anxiety Level of Children During Anesthesia Induction - A Randomized Controlled Trial
Brief Title: Effect of Parental Presence on Anxiety of Children During Induction of Anesthesia
Acronym: PPIA
Status: Completed | Type: Observational
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Ghulam Fatima, Principal Investigator, Liaquat National Hospital & Medical College
Other Study IDs: LNHMC karachi; Dr ghulam fatima (Other: liaquat national hospital)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Preoperative Anxiety
Keywords: Pre-operative anxiety,; Minor surgery,; parental presence during induction of anesthesia; modified Yale Preoperative Anxiety Scale
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 35 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPIA: children anesthetized in the presence of parents: PPIA: Children induced during the presence parents to assess the level of anxiety while aneshetizing.
- Control group: Control Group: children induced without the parental presence to assess level of anxiety during anesthitizing.

SUMMARY:
Anxiety is when children feel scared, worried, or nervous before or during anesthesia induction. This can happen because they don't know what's happening, are scared of the hospital or medical equipment, or are worried about being separated from their parents.

When parents are present, they can:

* Provide emotional support and reassurance
* Distract the child from scary things
* Help the child feel more calm and safe This can help reduce the child's anxiety levels.

When parents are not present, children may feel:

* More scared and anxious
* Alone and unsupported
* More worried about what's happening This can increase the child's anxiety levels. we can prepare children and parents beforehand about what will happen
* Allow parents to be present during anesthesia induction
* Use distraction techniques like toys or videos
* Use gentle and calm anesthesia induction techniques By doing these things, we can help reduce anxiety in children and make the experience less scary for them.

DETAILED DESCRIPTION:
Induction of pediatric anesthesia represents a highly stressful event for children, often resulting in preoperative anxiety that can impair the child's perioperative experience and result in adverse postoperative outcomes. It has been proposed that parental presence during induction of anesthesia Preoperative anxiety is linked to postoperative maladaptive behaviors, such as pain following surgery, insomnia, conflicts between the child and his parent, separation anxiety, increased urinary frequency during the night, reduced appetite, lack of interest, agitation, and alienation.may be a non-pharmacologic intervention to reduce children's anxiety. In patients with extreme anxiety, unfavorable postoperative behaviors after anesthesia induction are likely to result in long-term issues, which adversely affect the process of recovery, and also develop a feeling of inadequate care. Parental presence at anesthesia induction is the interaction that takes place in the induction room during the course of anesthesia induction between the child, parent, anesthesiologist, and perioperative nurses.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients
* aged 5-10 years
* minor surgery
* duration <1 hour
* ASA 1 and ASA 2 patients

Exclusion Criteria:

* Patients and attendant refusal
* Emergency surgeris
* Renal insuffciency
* Age less than 5 and more than 10 years

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A group of patients selected from a surgical day care units and wards who presented for minor elective surgical procedures.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Anxiety | minimum 2 to 3 minutes during Induction of anesthesia
  Modified yale preoperative anxiety scale (myPAS) assess activity, vocaliztion and Emotional expressivity andstate of apparent arousal. score 4 to 18 4 means no anxiety and 18 means highly anxious

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima Dr Ghulam Fatima, Principal Investigator — Liaquat National Hospital and Medical College
Locations (1):
- Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
1. *Patient confidentiality*: Sharing IPD could compromise patient confidentiality and anonymity, potentially harming participants or their families.
  2. *Sponsor's intellectual property*: Clinical trial sponsors may consider IPD as their intellectual property, and sharing it could compromise their commercial interests.
  3. *Competitive advantage*: Sharing IPD could provide competitors with valuable insights, potentially eroding the sponsor's competitive advantage.
     Data quality and validation*: IPD may require additional validation and quality control checks before sharing, which can be time-consuming and resource-intensive.
  4. *Methodological limitations*: Sharing IPD without proper context and methodology information may lead to misinterpretation or misuse of the data.
  5. Informed consent*: Participants may not have provided informed consent for their data to be shared, which could raise ethical concerns.

REFERENCES:
- See also: Fraley B. Preoperative anxiety and education in the adolescent population. Beckley, West Virginia: Mountain State University; 2007. 2. Caumo W, Ferreira MBC. Perioperative anxiety: psychobiology and effects in postoperative recovery. The Pain Clinic. 201 — https://pdfs.semanticscholar.org/e9d8/cf809a6ba7e2b96f84ea67f8bfbc7d058422.pdf